CLINICAL TRIAL: NCT05527678
Title: Assessment of Quality of Life in Patients Who Participated in the Promorea 1 Study
Brief Title: 5 Years Quality of Life and Early Mobilization in ICU
Acronym: Promorea-qol
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: CHRO-2022-02
Record Dates: First submitted 2022-08-30; First posted 2022-09-02 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Quality of Life; ICU Acquired Weakness; Morality
Keywords: ICU; Quality of life; Medical research council sum score; Mortality; early mobilization
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 5 years ICU survivors: Survivors 5 years after ICU and who participated in the Promorea1 study will be contacted to assess their quality of life.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Written or by phone

SUMMARY:
In a study published in 2018 the research team had collected the Medical Research Council score (MRCs) at Intensive Care Unit (ICU) discharge.

The investigators would like to be able to examine, if the preliminary results obtained by in 2020 by Van Aerde's team are confirmed in their cohort.

The investigators hypothesize that patients with an MRCs less than or equal to 55 at discharge from the ICU, have a higher mortality rate than those with a score greater than 55.

The investigators would also like to examine whether or not an MRCs score ≤ 55 is associated with a difference in quality of life and autonomy, after 5 and more years post ICU.

DETAILED DESCRIPTION:
Study design Prospective, observational study.

1. Research of vital status
2. Completion of two questionnaires (Short Form-36 and Katz Index of Independence in Activities of Daily Living), to assess quality of life and level of autonomy in activities of daily living, either by telephone or completed directly by hand by the patient from his place of residence.

ELIGIBILITY:
Inclusion Criteria:

* Have participated in the Promorea1 study
* Alive at the time the questionnaires were sent

Exclusion Criteria:

* Opposition to the use of vital status data
* Extra-national patient not on the national registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who participated in the PROMOREA 1 study, whose vital status is "alive" at least 5 years after their discharge from the ICU (INSEE file, MatchID search engine, https://deces.matchid.io/search?fuzzy=false), will be recontacted by mail at the last known address and by phone at the last known number if they do not answer the mail.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
5 years mortality | Before sending questionnaires
  Vital status

SECONDARY OUTCOMES:
Medical Outcomes Study 36-item Short-Form Health Survey | through study completion, an average of 6 months
  The 36-Item Short Form Survey (SF-36) is an oft-used, well-researched, self-reported measure of health. It stems from a study called the Medical Outcomes Study.
  It comprises 36 questions which cover eight domains of health.
  The recommended scoring system for the SF-36 is a weighted Likert system for each item. Items in the subscales are summed to obtain a summary score for each subscale or dimension. Each of the 8 summary scores is linearly transformed on a scale from 0 (negative to health) to 100 (favorable to health) to obtain a score for each subscale.
Katz Index of Independence in Activities of Daily Living questionnaire | through study completion, an average of 6 months
  The Katz Index of Independence in Activities of Daily Living, commonly referred to as the Katz ADL, is the most appropriate instrument to assess functional status as a measurement of the client's ability to perform activities of daily living independently. Clinicians typically use the tool to detect problems in performing activities of daily living and to plan care accordingly. The Index ranks adequacy of performance in the six functions of bathing, dressing, toileting, transferring, continence, and feeding. Clients are scored yes/no for independence in each of the six functions.
  A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment.
  The instrument is most effectively used among older adults in a variety of care settings, when baseline measurements, taken when the client is well, are compared to periodic or subsequent measures.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume FOSSAT, Pt Msc, Principal Investigator — Centre Hospitalier Régional d'Orléans
Locations (1):
- Centre Hospitalier Régional d'Orléans, Orléans, Centre-Val de Loire, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Result] Fossat G, Baudin F, Courtes L, Bobet S, Dupont A, Bretagnol A, Benzekri-Lefevre D, Kamel T, Muller G, Bercault N, Barbier F, Runge I, Nay MA, Skarzynski M, Mathonnet A, Boulain T. Effect of In-Bed Leg Cycling and Electrical Stimulation of the Quadriceps on Global Muscle Strength in Critically Ill Adults: A Randomized Clinical Trial. JAMA. 2018 Jul 24;320(4):368-378. doi: 10.1001/jama.2018.9592. PMID 30043066
- [Result] Van Aerde N, Meersseman P, Debaveye Y, Wilmer A, Gunst J, Casaer MP, Bruyninckx F, Wouters PJ, Gosselink R, Van den Berghe G, Hermans G. Five-year impact of ICU-acquired neuromuscular complications: a prospective, observational study. Intensive Care Med. 2020 Jun;46(6):1184-1193. doi: 10.1007/s00134-020-05927-5. Epub 2020 Jan 22. PMID 31970446